CLINICAL TRIAL: NCT05154331
Title: Antenatal and Postnatal Care Research Collective - Household Survey (ARCH)
Acronym: ARCH
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Zambia (Other)
Responsible Party: Sponsor
Other Study IDs: 21-1370
Record Dates: First submitted 2021-11-29; First posted 2021-12-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Maternal Health; Pregnancy Outcomes
Keywords: pregnancy health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women of reproductive age: Women 15-49 years of age

SUMMARY:
The overarching goal of the ARCH Survey is to establish a prospective longitudinal pregnancy surveillance study in Lusaka, Zambia, to precisely characterize the pregnancy rate and outcomes of women of reproductive age prior to, during, and following pregnancy and to investigate the structural, sociodemographic, and clinical covariates that contribute to adverse outcomes in each reproductive epoch.

DETAILED DESCRIPTION:
The overall purpose of this study is to better understand the health and well-being of women before and after they become pregnant and of their infants. This information will contribute to the understanding of the health needs of women and their children, which may help doctors provide mothers and children with better care in the future.

Participants in this study will be visited four times a year (every 3 months) for up to three years in total. At each visit a review of their medical records, a brief physical exam and urine pregnancy test will be conducted. Participants will also answer survey questions and self-collect vaginal swabs for future testing. We will enroll up to 5,500 women and include any infants that are born to them during their study participation.

ELIGIBILITY:
We will initially obtain verbal consent from the head of household (HoH), defined as an available adult (> 18 years old) who is able to provide information about household composition for pre-screening purposes. We will then identify potentially eligible women of reproductive age within each household and invite them to complete study screening procedures.

Women of reproductive age eligibility criteria

Inclusion criteria:

* Verbal consent obtained from head-of-household
* 15-49 years of age and a member of household in the catchment area
* Willing and able to provide written informed consent or assent with next-of-kin consent
* Willing to undergo study procedures

Exclusion criteria:

Any other condition (social or medical) that, in the opinion of the study staff, would make participation unsafe or complicate data interpretation. Study staff may note physical, psychological, or social conditions not explicitly stated in the eligibility criteria that could make some women poor candidates for study participation.

Ages: 1 Day to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women of reproductive age and their infants born during their study participation
Sampling Method: Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cohort Pregnancy Ratio | enrollment - 36 months
  Defined as the total number of pregnancies, including live births, stillbirths, and abortions per 1000 women aged 15-49.
Cohort Term Live Birth Ratio | enrollment - 36 months
  Defined as the proportion of pregnancies that result in a live birth at or beyond 37 gestational weeks per 1,000 pregnancies.
Cohort Infant Mortality Ratio | enrollment - 36 months
  Defined as the number of deaths in children under one year of age per 1,000 live births.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Stringer, Principal Investigator — University of North Carolina, Chapel Hill; Wilbroad Mutale, MD, Principal Investigator — University of Zambia (UNZA) Lusaka, Zambia
Locations (1):
- University of Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9-36 months following publication
Access Criteria: noted above